CLINICAL TRIAL: NCT01387932
Title: Phase 3 Prospective, Randomized, Blinded, and Controlled Investigation of HepaSphere/QuadraSphere Microspheres for Delivery of Doxorubicin for the Treatment of Hepatocellular Carcinoma
Brief Title: HepaSphere/Quadrasphere Microspheres for Delivery of Doxorubicin for the Treatment of Hepatocellular Cancer
Acronym: HiQuality
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The clinical study was terminated due to the inability to meet target enrollment.
Sponsor: Merit Medical Systems, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HCC-P3-11-01
Record Dates: First submitted 2011-04-11; First posted 2011-07-06 (Estimated); Results first posted 2021-11-30 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-11

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular carcinoma; TACE; HepaSphere Microspheres; QuadraSphere Microspheres; Doxorubicin
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Desmoglein 3; Ethiodized Oil; Doxorubicin

STUDY DESIGN:
Intervention Model Description: Participants are randomized 1:1 to receive either 1. A Conventional TACE (Trans Arterial Chemoembolization) procedure using PVA, lipiodol and doxorubicin (cTACE), or 2. HepaSphere/QuadraSphere Microspheres loaded with doxorubicin for Trans Arterial Chemoembolization (hqTACE). Participants in both treatment arms will be followed for overall survival, the primary study endpoint.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants are blinded to the treatment they are randomized to (cTACE or hqTACE). Central Reviewers (two interventional radiologists) will evaluate study participant's liver MRIs to assess the tumor response. The Central Reviewers will be blinded to the treatment the participant received.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: Yes

ARMS (2):
- HepaSphere/QuadraSphere TACE (Experimental): HepaSphere/QuadraSphere TACE
  Interventions: Device: HepaSphere/QuadraSphere Microspheres
- Conventional TACE (Active Comparator): Conventional TACE
  Interventions: Procedure: PVA, lipiodol, doxorubicin

INTERVENTIONS:
Device: HepaSphere/QuadraSphere Microspheres — HepaSphere/QuadraSphere Microspheres loaded with doxorubicin
  Arms: HepaSphere/QuadraSphere TACE
Procedure: PVA, lipiodol, doxorubicin — Conventional TACE procedure using PVA, lipiodol and doxorubicin
  Arms: Conventional TACE

SUMMARY:
The purpose of this study is to evaluate overall survival in patients diagnosed with hepatocellular cancer (HCC) treated with HepaSphere/QuadraSphere Microspheres loaded with chemotherapeutic agent doxorubicin compared to conventional transarterial chemoembolization with particle PVA, lipiodol, and doxorubicin.

DETAILED DESCRIPTION:
This phase three, interventional, and prospective study consists of a patient population that has advanced liver cancer (hepatocellular cancer [HCC]) that cannot be removed by standard therapies such as surgical removal, liver transplant, and/or ablation.

Embolics and drug eluting embolics are being used by interventional radiologists to try and shrink or kill the tumor area.

Patients that met eligibility criteria, wanted to participate in the study, and signed the informed consent form (ICF) made up the study subject population. Subjects were randomized on a 1:1 basis (subjects were blinded to arm they were randomized to).

Post randomization and within four weeks of the first chemoembolization procedure all subjects had a baseline MRI. Following, the first chemoembolization procedure (hqTACE or cTACE) or 'cycle' was completed. Subjects can (per protocol) receive up to 3 TACE cycles. Within 4 weeks after any TACE cycle, an MRI and labs should be conducted/collected to evaluate disease status (reduction vs progression) and measure treated lesions. Any residual disease that is present after after the first TACE will undergo the next TACE cycle (maximum of three). However, if the liver MRI shows a complete response (absence of HCC) then no additional TACE procedures are performed and the subject is followed for survival.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following inclusion criteria in order to be entered into the study:

1. Age 18 or older
2. Patient has signed informed consent
3. Patient must have a diagnosis of hepatocellular cancer confirmed by at least one of the following:

i. Histological confirmation ii. Magnetic resonance imaging (MRI) result with early enhancement and delayed enhancement washout of at least one solid liver lesion > 1 cm. Patient must also have evidence of cirrhosis or have chronic hepatitis B.

iii. Contrast enhanced computed tomography (CT) with early enhancement and delayed enhancement washout of at least one solid liver lesion > 1cm. Patient must also have evidence of cirrhosis or have chronic hepatitis B.

d. Patient must not be suitable for treatment by resection or percutaneous ablation at time of study entry.

Patients not suitable for ablation due to lesion location may be enrolled

e. Patient MUST meet at least ONE of the following criteria:

i. Stage Child-Pugh B 7 ii. Recurrent HCC iii.Performance status ECOG 1

f. Patient has a life expectancy of at least 6 months

g. Absence of occlusive thrombus to the main portal trunk

Exclusion Criteria:

If patients meet any of the following criteria they may not be entered into the study:

1. Current or previous treatment with chemo- or radiation therapy or sorafenib
2. Previous treatment with any form of transarterial embolization for HCC
3. Patients with current or history of any other cancer except non-melanomatous skin cancer
4. Female patients who are pregnant, breastfeeding, or premenopausal and not using an effective method of contraceptive
5. Performance status ECOG > 2
6. Child-Pugh scores >7
7. Active gastrointestinal bleeding
8. Evidence of uncorrectable bleeding diathesis
9. Extra-hepatic spread of the HCC
10. Total Bilirubin > 3 mg/dL
11. >50% tumor involvement of the liver
12. Infiltrative or diffuse HCC
13. Encephalopathy not adequately controlled medically
14. Presence of ascites not controlled medically
15. Presence of medically relevant localized or systemic infection, other than hepatitis B, C, D, E or G
16. Any contraindication for MRI (eg. metallic implants)
17. Allergy to contrast media that cannot be managed with prophylaxis
18. Allergy to iodized oil
19. Any contraindication to arteriography
20. Any contraindication for doxorubicin administration, including the following:

i. White Blood Cell count (WBC) <3000 cells/mm₃

ii. Absolute Neutrophil <1500 cells/mm₃

iii. Cardiac ejection fraction <50%

iv. Other condition deemed exclusionary by physician

u. Any contraindication for hepatic embolization, including the following:

i. Porto-systemic shunt, or an arteriovenous shunt that cannot be adequately closed prior to chemoembolization

ii. Hepatofugal blood flow

iii. Serum creatinine > 2mg/dL

iv. Uncorrectable impaired clotting

1. Platelet <50,000/mm₃
2. International Normalized Ratio (INR) > 1.4
3. Activated Prothrombin Time (aPTT) less than 21 or greater than 40

   v. AST > 5X upper limit of normal for lab

   vi. ALT > 5X upper limit of normal for lab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 235 (Actual)
Dates: Start 2011-06 (Actual); Primary Completion 2021-02 (Actual); Study Completion 2021-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Soulen, MD, Principal Investigator — University of Pennsylvania; Riccardo Lencioni, MD, Study Chair — Independent Radiology Panel; Josep Llovet, MD, Study Chair — Data Safety Monitoring Board
Locations (23):
- United States (18):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Tuscon Medical Center, Tucson, Arizona
  - Greater Arkansas Veterans Healthcare, Little Rock, Arkansas
  - VA Greater Los Angeles Healthcare System, Los Angeles, California
  - UCLA, Los Angeles, California
  - Palo Alto Veterans Institute for Research, Palo Alto, California
  - Stanford University, Stanford, California
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - Tampa General Hospital, Tampa, Florida
  - Northwestern University, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Albany Medical Center, Albany, New York
  - Mount Sinai Medical Center, New York, New York
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Albert Einstein Healthcare, Philadelphia, Pennsylvania
  - VA Pittsburgh Healthcare System, Pittsburgh, Pennsylvania
  - MUSC Medical Center (Medical University of South Carolina), Charleston, South Carolina
  - UT Health and Science Center, San Antonio, Texas
- University Hospitals K.U. Leuven (Dept of Hematology), Leuven, Belgium
- France (2):
  - Hospital Saint Andre, Bordeaux
  - Hospital Paul Brousse, Villejuif
- Evgenidion University Hospital, Athens, Greece
- S. Croce e Carle Hospital, Cuneo, Italy

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study enrollment began in June 2011 and ended in May 2017.
Pre-assignment Details: Of the 235 subjects that were randomized, 224 were treated. Eleven (11) randomized subjects did not receive treatment, 5 of which were not treated at the investigators discretion and 6 that withdrew consent.
Groups:
- HepaSphere/QuadraSphere TACE: HepaSphere/QuadraSphere TACE
  Transarterial chemoembolization in participants with localized, non-resectable hepatocellular carcinoma utilizing HepaSphere/QuadraSphere Microspheres loaded with doxorubicin.
- Conventional TACE: Conventional TACE
  Transarterial chemoembolization in participants with localized, non-resectable hepatocellular carcinoma utilizing PVA, lipiodol, doxorubicin.
Period: Randomized and Treated
Arm/Group | HepaSphere/QuadraSphere TACE | Conventional TACE
Started | 118 | 117
Completed | 111 | 113
Not Completed | 7 | 4
Not completed — Physician Decision | 3 | 2
Not completed — Withdrawal by Subject | 4 | 2
Period: Completion of TACE Cycle
Arm/Group | HepaSphere/QuadraSphere TACE | Conventional TACE
Started | 111 | 113
Completed (One hundred percent of the hqTACE arm and 100% of the cTACE arm received their first TACE Cycle.) | 111 | 113
Not Completed | 0 | 0
Period: Survival Follow-up
Arm/Group | HepaSphere/QuadraSphere TACE | Conventional TACE
Started (All subjects that completed at least one TACE cycle were eligible for long-term survival follow-up.) | 111 | 113
Completed | 27 | 23
Not Completed | 84 | 90
Not completed — Liver Transplant | 24 | 28
Not completed — Additional treatment excluding liver transplant | 52 | 53
Not completed — Withdrawal by Subject | 2 | 4
Not completed — Lost to Follow-up | 6 | 5

BASELINE CHARACTERISTICS:
Population: Baseline Analysis Population are the number of subjects that were randomized to that study arm.
Groups:
- Total: Total of all reporting groups
Arm/Group | HepaSphere/QuadraSphere TACE | Conventional TACE | Total
Number analyzed (Participants) | 118 | 117 | 235
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.0 (8.95) | 64.2 (8.40) | 64.1 (8.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 20 | 44
  Male | 94 | 97 | 191
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  RACE (NIH/OMB): Asian | 8 | 6 | 14
  RACE (NIH/OMB): Native Hawaiian or Pacific Islander | 0 | 1 | 1
  RACE (NIH/OMB): Black or African American | 8 | 9 | 17
  RACE (NIH/OMB): White | 95 | 96 | 191
  RACE (NIH/OMB): More than one race | 2 | 1 | 3
  RACE (NIH/OMB): Unknown or Not Reported | 5 | 4 | 9
Region of Enrollment [Count of Participants; unit: Participants] — Population: The Analysis Population is the 224 treated subjects and not the 235 randomized subjects, as the 11 subjects either withdrew consent or did not receive any study treatments as they were deemed ineligible by the treating investigator.
  Participants
    Greece: number analyzed (Participants) | 111 | 113 | 224
    Greece | 25 | 24 | 49
    Belgium: number analyzed (Participants) | 111 | 113 | 224
    Belgium | 2 | 2 | 4
    United States: number analyzed (Participants) | 111 | 113 | 224
    United States | 78 | 79 | 157
    Italy: number analyzed (Participants) | 111 | 113 | 224
    Italy | 4 | 4 | 8
    France: number analyzed (Participants) | 111 | 113 | 224
    France | 2 | 4 | 6

OUTCOME MEASURES:

1. Primary Outcome: Median Overall Survival
Description: Median overall survival will be calculated using the Intent-to-Treat (ITT) population in each treatment arm when the last subject has completed two years of follow up after their first study TACE procedure. Per protocol, study subjects were followed for survival until death or deemed lost to follow up. All deaths are reported within safety.
Time Frame: 2 years
Population: The analysis populations for both the HepaSphere/QuadraSphere TACE (hqTACE) and conventional TACE (cTACE) arms included all subjects with HCC that received one or more protocol specified TACE procedures.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | HepaSphere/QuadraSphere TACE | Conventional TACE
Number analyzed (Participants) | 27 | 23
Months | 9.0 [8.02 to 9.99] | 7.0 [3.39 to 10.61]

2. Secondary Outcome: Objective Response Rates (ORR)
Description: The Objective Response Rate will be calculated for the ITT population by adding the number of participants that were determined to have complete or partial response (utilizing mRECIST criteria) and dividing by the number of ITT participants.
Time Frame: Study was terminated early so analysis of additional outcome(s) were not possible.
Population: Data was not collected.
Arm/Group | HepaSphere/QuadraSphere TACE | Conventional TACE
Number analyzed (Participants) | 0 | 0

3. Other Pre Specified Outcome: Number of TACE-Related Adverse Events in Subjects Treated With HepaSphere/QuadraSphere vs Subjects Treated With Conventional TACE.
Description: The number of TACE- Related adverse events experienced by subjects treated with HepaSphere/QuadraSphere will be compared to the number of TACE-related adverse events experienced by subjects treated with conventional TACE.
  Adverse events were recorded for treated subjects from the date of randomization up to and including 30 days post the last study MRI.
Time Frame: 30 days
Population: Analysis populations were: 1. All subjects treated with HepaSphere/QuadraSphere TACE and 2. All subjects treated with conventional TACE.
Measure: Number; unit: A TACE related Adverse Event
Arm/Group | HepaSphere/QuadraSphere TACE | Conventional TACE
Number analyzed (Participants) | 111 | 113
A TACE related Adverse Event | 149 | 164

ADVERSE EVENTS:
Time Frame: All adverse events (AEs) occurring between the date of randomization until study termination, an average of 25.8 and 28.0 months per participant in the hqTACE and cTACE arms respectively.
Arm/Group | HepaSphere/QuadraSphere TACE | Conventional TACE
All-Cause Mortality (participants affected / at risk) | 100/111 | 93/113
Serious Adverse Events (participants affected / at risk) | 23/111 | 21/113
Other Adverse Events (participants affected / at risk) | 86/111 | 87/113
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HepaSphere/QuadraSphere TACE (N=111) | Conventional TACE (N=113)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (2) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 5 (6)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal ulcer hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus paralytic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mesenteric vein thrombosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal varices hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Varices oesophageal (Gastrointestinal disorders) | 1 (1) | 0 (0)
Multi-organ failure (General disorders) | 0 (0) | 2 (2)
Pain (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic infarction (Hepatobiliary disorders) | 0 (0) | 1 (1)
Portal vein thrombosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Bacterial infection (Infections and infestations) | 1 (1) | 0 (0)
Enterococcal bacteremia (Infections and infestations) | 0 (0) | 1 (1)
Groin abscess (Infections and infestations) | 1 (1) | 0 (0)
Lobar pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Peritonitis bacteria (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 2 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post embolisation syndrome (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1)
Blood glucose increased (Investigations) | 0 (0) | 1 (1)
Body temperature increased (Investigations) | 1 (1) | 0 (0)
Liver function test abnormal (Investigations) | 0 (0) | 2 (4)
Food intolerance (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Hepatic encephalopathy (Nervous system disorders) | 0 (0) | 2 (3)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (3) | 1 (2)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 2 (2)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HepaSphere/QuadraSphere TACE (N=111) | Conventional TACE (N=113)
Abdominal pain (Gastrointestinal disorders) | 27 (40) | 30 (40)
Abdominal pain upper (Gastrointestinal disorders) | 17 (22) | 16 (20)
Ascites (Gastrointestinal disorders) | 7 (9) | 5 (7)
Constipation (Gastrointestinal disorders) | 11 (14) | 13 (14)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 10 (12)
Nausea (Gastrointestinal disorders) | 33 (48) | 32 (45)
Vomiting (Gastrointestinal disorders) | 10 (16) | 12 (16)
Catheter site pain (General disorders) | 6 (7) | 4 (4)
Chills (General disorders) | 2 (3) | 6 (7)
Fatigue (General disorders) | 23 (26) | 24 (25)
Oedema peripheral (General disorders) | 4 (5) | 7 (7)
Pyrexia (General disorders) | 21 (32) | 19 (20)
Post embolisation syndrome (Injury, poisoning and procedural complications) | 21 (39) | 21 (38)
Alanine aminotransferase increased (Investigations) | 12 (16) | 9 (11)
Alpha 1 foetoprotein increased (Investigations) | 7 (7) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 12 (15) | 10 (14)
Blood alkaline phosphatase increased (Investigations) | 8 (10) | 4 (6)
Blood bilirubin increased (Investigations) | 8 (8) | 4 (4)
Weight decreased (Investigations) | 9 (10) | 9 (9)
Decreased appetite (Metabolism and nutrition disorders) | 6 (8) | 17 (18)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (6) | 8 (8)
Headache (Nervous system disorders) | 6 (6) | 3 (3)
Insomnia (Psychiatric disorders) | 6 (6) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 6 (6)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 22 (22)

LIMITATIONS AND CAVEATS:
Study was terminated early due to insufficient enrolment to support analysis of endpoints. A full safety analysis was completed and is reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-04-21): https://cdn.clinicaltrials.gov/large-docs/32/NCT01387932/Prot_SAP_000.pdf